CLINICAL TRIAL: NCT04019717
Title: A Phase 2 Study Assessing the Safety and Efficacy of AT-527 in Combination With Daclatasvir in Subjects With Chronic HCV Infection
Brief Title: Study of AT-527 in Combination With Daclatasvir in Subjects With Hepatitis C Virus (HCV) Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT-01B-002; 2019-001431-31 (EudraCT Number)
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-05

CONDITIONS: Hepatitis C; Hepatitis C, Chronic; Chronic Hepatitis C; Hepatitis C Virus Infection; HCV Infection
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — AT-511; daclatasvir

STUDY DESIGN:
Intervention Model Description: Subjects will receive 8 or 12 weeks of treatment, based on treatment response.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8 weeks (Experimental)
  Interventions: Drug: AT-527; Drug: Daclatasvir
- 12 weeks (Experimental)
  Interventions: Drug: AT-527; Drug: Daclatasvir

INTERVENTIONS:
Drug: AT-527 — Nucleotide prodrug inhibitor of HCV nonstructural protein 5B (NS5B) polymerase
Drug: Daclatasvir — Inhibitor of HCV nonstructural protein 5A (NS5A)

SUMMARY:
The study will assess the safety and efficacy of AT-527 in combination with daclatasvir after 8 or 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 18-35 kg/m2
* Must agree to use protocol-specified methods of contraception
* Negative pregnancy test
* HCV genotype 1
* Documented history compatible with chronic hepatitis C
* HCV RNA ≥ 10,000 IU/mL at Screening.
* Willing to comply with the study requirements and to provide written informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Infected with hepatitis B virus or HIV
* Abuse of alcohol or drugs
* Prior exposure to any HCV NS5A inhibitor
* Cirrhosis
* Use of other investigational drugs within 30 days of dosing
* Other clinically significant medical conditions or contraindications to daclatasvir

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving sustained virologic response (SVR) | 12 weeks after end of treatment
  SVR defined as the HCV RNA < lower limit of quantitation (LLOQ) at 12 weeks after end of treatment
Incidence of treatment-emergent adverse events | Through 4 weeks after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jian Zhou, PhD, Study Director — Atea Pharmaceuticals, Inc.
Locations (3):
- Clinical Trial Site, Antwerp, Belgium
- Clinical Trial Site, Phoenix, Mauritius
- Clinical Trial Site, Chisinau, Moldova